CLINICAL TRIAL: NCT06926413
Title: An Open-label, Fixed-sequence Phase I Clinical Study Evaluating the Effect of Multiple Oral Doses of Aumolertinib on the Pharmacokinetics of Midazolam in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study Evaluating the Effect of Aumolertinib on the Pharmacokinetics of Midazolam in Patients With NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10296-109
Record Dates: First submitted 2025-03-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10296 (Experimental)
  Interventions: Drug: Aumolertinib；midazolam

INTERVENTIONS:
Drug: Aumolertinib；midazolam — Midazolam :
  The enrolled subjects will receive a single oral dose of Midazolam 2 mg (2 mg/mL, 1 mL) on D1 of the run-in period and on C2D1.
  Aumolertinib :
  Starting from C1D1, the enrolled subjects will receive oral dose of aumolertinib 110 mg (55 mg/tablet, 2 tablets) once daily until the criteria for terminating treatment are met.

SUMMARY:
This is an open-label, fixed-sequence Phase I clinical study that evaluates the effect of multiple doses of aumolertinib on the pharmacokinetics of midazolam (CYP 3A4 probe substrate) in sensitive EGFR (Epidermal Growth Factor Receptor) mutation-harboring patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence Phase I clinical study that evaluates the effect of multiple doses of aumolertinib on the pharmacokinetics of midazolam (CYP 3A4 probe substrate) in sensitive EGFR (Epidermal Growth Factor Receptor) mutation-harboring patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).

The study includes D1 (Day 1)-D2 (Day 2) of run-in period, C1D1 (Cycle 1 Day 1)-C1D21 (Cycle 1 Day 21) and C2D1 (Cycle 2 Day 1)-C2D2 (Cycle 2 Day 2). The enrolled subjects will receive a single oral dose of midazolam 2 mg (2 mg/mL, 1 mL) on D1 of the run-in period and on C2D1; and receive oral dose of aumolertinib 110 mg (55 mg/tablet, 2 tablets) once daily from C1D1 to C2D2.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant should sign an informed consent form before the trial. 2. Male or female age≥18 years, at the time of signing the informed consent. 3. Histologically or cytological confirmation diagnosis of locally advanced or metastatic (IIIB/IIIC/IV) NSCLC; 4. Participant must fulfill one of below:

  1. Participants who have not received any prior anti-tumor systemic therapy, and the tumor must harbor at least one of the EGFR mutations (ex19del or L858R, single mutation or combined with other EGFR mutations are both acceptable).
  2. Participant who received first-generation EGFR-TKI in the locally advanced or metastatic setting and have documented radiological progression prior to enrolling in the study, and the tumor must harbor EGFR T790M mutation.

     5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1 and no deterioration in the previous two weeks with a minimum life expectancy of 12 weeks.

     6. Male or female should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and female should not breastfeed.

     Exclusion Criteria:
* 1. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study intervention with the exception of alopecia and Grade 2 neurotoxicity related to prior platinum-therapy.

  2. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least four weeks prior to start of study intervention.

  3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding within two weeks prior to the first dose of study intervention, active infection (e.g., active HBV infection, HCV infection), or HIV infection, which in the Investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardise compliance with the protocol.

  4. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.

  5. Refractory nausea, vomiting, or chronic GI disorders; Participants unable to swallow oral medication or participants with GI disorders or significant GI resection likely to interfere with the absorption of study intervention.

  6. Participant has any disease or condition that, in the judgment of the physician, may increase the risk to the safety or interfering with study assessments.

  7. Participant with a known hypersensitivity to study intervention (Aumolertinib and Midazolam), structural analog, or any of the excipients of the products.

  8. Past medical history of ventilation difficulties or severe sleep apnea syndrome.

  9. Patient with acute angle-closure glaucoma or untreated open-angle glaucoma. 10. Patient which in the Investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardise compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cmax, of midazolam and 1-hydroxymidazolam (midazolam combined with aumolertinib/midazolam administrated alone) | Day 1
  Maximum plasma concentration
AUC0-t of midazolam and 1-hydroxymidazolam (midazolam combined with aumolertinib/midazolam administrated alone) | Day 1
  Area under the plasma concentration-time curve from 0-t
AUC0-∞ of midazolam and 1-hydroxymidazolam (midazolam combined with aumolertinib/midazolam administrated alone) | Day 1
  Area under the plasma concentration-time curve from 0-∞

SECONDARY OUTCOMES:
Cmin of aumolertinib, HAS-719 and other major metabolites (if applicable) | Day 1
  Minimum plasma concentration
Cmax of aumolertinib, HAS-719 and other major metabolites (if applicable) | Day 1
  Maximum plasma concentration
AUC0-24h of aumolertinib, HAS-719 and other major metabolites (if applicable) | Day 1
  Area under the plasma concentration-time curve from 0-24h
Tmax of aumolertinib, HAS-719 and other major metabolites (if applicable) | Day 1
  Time to reach Cmax
Incidence and severity of adverse event | D25

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of the First Addiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China